CLINICAL TRIAL: NCT06637709
Title: Persistent Pain in Pharmacologically or Surgical Treated Osteoarthritis: the Role of the Mu-Lympho Marker As a Candidate Innovative Diagnostic Tool
Brief Title: Persistent Pain in Pharmacologically or Surgical Treated Osteoarthritis: Role of Mu-Limpho Marker
Acronym: MLM
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 22/23
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain; Osteo Arthritis Knee
Keywords: pain biomarkers; Mu opioid receptor; tailored therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: patients with symptomatic knee osteoarthritis (OA): Experimental group includes a subgroup: OA patients from the experimental group requiring primary TKA due to the failure of conservative treatment, thus undergoing surgical intervention.
- Control group: subjects without any chronic pain: subjects undergoing occupational health surveillance matched by age, sex and psychological profile with the experimental group patients

SUMMARY:
The goal of this prospective observational study is to analyze the percentage of expression of B and NK cells expressing Mu opioid receptor on their surface, named Mu-Lympho-Marker (MLM), to measure pain progression in Osteoarthritis patients and its association with specific rehabilitation programs. In particular, we want to analyze the role of MLM as diagnostic biomarker of pain chronicization.

The main aims are:

* to explore the relationship between Mu+ B and NK cells percentage and pain progression in OA patients, also investigating whether this characteristic is associated to particular outcome of pharmacological and/or surgery interventions and rehabilitation
* to characterize Mu+ B and NK cells in terms of maturation states, activation/inhibition and functional properties, as well as their ability to respond to Mu stimulation, in order to understand whether these cells can have a role in the pathogenesis of OA associated CP
* to investigate the potential confounding effect of other biological and psychological elements in the relationship between the MLM and OA pain progression

Researchers will compare two study groups:

1. Experimental group: subjects suffering from symptomatic knee OA. 1S)surgical subgroup: OA patients from the experimental group requiring primary TKA due to the failure of conservative treatment, thus undergoing surgical intervention;
2. Control group: subjects without any chronic pain, undergoing occupational health surveillance matched by age, sex and psychological profile with the experimental group patients Participants will be asked to do blood sample collections at specific time points to evaluate MLM stability over time and its modulation according to pharmacological/surgical and rehabilitation interventions. Subjects in the control group will undergo 2 blood sample collections. Pain assessment will be performed at all scheduled time points to correlate pain severity with Mu expression in B and NK cells.

DETAILED DESCRIPTION:
All patients will undergo the blood sampling at the day of the enrollment (T0), at 1 month (T1), 3 months (T2) and 6 months(T3) after the enrollment. The subgroup of patients requiring primary TKA will undergo blood sampling the day of the surgical intervention (T1-S), the 5th day (T2-S), and the 90th day after the intervention (T3-S). Pain-free subjects will undergo blood sampling the day of the enrollment (T0) and 6 months (T3) later.

Participants will be asked to self-fill the 11-point numerical rating scale (NRS) test, where 0= No pain and 10= worst possible pain, 2) the Italian version of the Brief Pain Inventory and the Italian version of the Neuropathic Pain Symptom Inventory NPSI (I-NPSI), 3) the Italian version of the Knee injury and Osteoarthritis Outcome Score (KOOS).

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis with disabling pain, age older than 18 years at the time of surgery, capability tocommunicate with healthcare professionals and give valid informed consent, and a willingness to participate in a 24-month follow-up.

Exclusion Criteria:

* (1) patients who underwent: surgical knee joint procedures; intra-articular knee injection in the last 3 months; (2) patients with: severe psychiatric disorder [excluding mild depression] or mental/cognitive impairment; a history [in the last 3 months] of fracture or trauma; (3) patients with a history in the last 6 months or currently suffering from: immunodeficiency diseases; connective tissue disease; infections; (4) pregnancy (5) patients ongoing opioids.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OA patients are referred to the Orthopedic and Traumatology Surgery Unit of the University Hospital Mater Domini (Catanzaro, Italy).
  The healthy subjects of the control group may be recruited not only from the Orthopedic and Traumatology Surgery Unit of the University Hospital Mater Domini but also from the IRCCS San Raffaele in Rome, during the corporate medical visit and from other approved studies.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Identification of differences in the percentage of Mu opioid receptor positive B and NK cells between experimental and control groups. | 3 years
  Characterization of Mu opioid receptor positive B/NK cells percentage of expression as a candidate biomarker for assessing the risk of pain persistency and chronicization following pharmacological, surgical, and/or rehabilitation interventions.

SECONDARY OUTCOMES:
Correlations between biological and psychological outcomes | 3 years
  The analysis of correlation between bilogical and psychological data will help to mitigate potential confounding effects and to optimized rehabilitation strategies based on study findings

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Roma, Roma, Roma, Italy